CLINICAL TRIAL: NCT04522271
Title: A Single Center, Randomized, Placebo-controlled, Double-blinded, Parallel, Pilot Clinical Trial to Assess Plant-derived Food-based Resistant Starches Individually Optimized for Patients With Crohn's Disease (CD) or Ulcerative Colitis (UC)
Brief Title: Resistant Starch in Pediatric Inflammatory Bowel Disease (Crohn's Disease or Ulcerative Colitis)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, David Mack, Director, CHEO IBD Centre, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20/04E
Record Dates: First submitted 2020-07-31; First posted 2020-08-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: Resistant Starch; Microbiome
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Resistant Starch

STUDY DESIGN:
Intervention Model Description: A single center, randomized, placebo-controlled, double-blinded, parallel, pilot clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinding will occur only if necessary to ensure study participants safety, interim analysis at 5 ± 1 months, or eligibility for our associated open label trial (OARS trial). Only Dr. Mack (Co-PI) can request to break the blind for safety reasons or eligibility for the OARS Trial; only Dr Stintzi (Co-PI) will request to break the blind for interim analysis. Once the blind is broken, the patient will be discontinued from study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Starch (Active Comparator): Once daily oral consumption of 7.5 g/m2 of an individually optimized resistant starch for approximately 5 months
  Interventions: Other: Resistant Starch
- Placebo (Placebo Comparator): Once daily oral consumption of a food-grade cornstarch that is readily digestible for approximately 5 months
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Resistant Starch — 7.5 g resistant starch/m2 oral consumption
  Arms: Resistant Starch
Other: Placebo — Placebo oral consumption of food-grade cornstarch
  Arms: Placebo

SUMMARY:
The purpose of the study is determine if a plant-based resistant starch that is optimized for the individual will target the underlying cause of inflammatory bowel disease and restore a "healthier" gut microbiome in pediatric participants with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent, or if appropriate, have an acceptable representative capable of giving consent on the participant's behalf.
* Enrolled in the main parent study.
* New ulcerative colitis diagnosis (mild/moderate) or Crohn's Disease diagnosis (moderate/severe) with colonic disease with or without terminal ileum disease, already started on oral corticosteroid or aminosalicylates for induction therapy at a time following diagnostic colonoscopy.
* Clinically responsive to induction medical therapy at enrollment (Crohn's Disease participants with a weighted pediatric Crohn's Disease activity index decrease of ≥ 17.5 points or ulcerative colitis participants with a pediatric ulcerative colitis activity index decrease of ≥ 15 points).
* Ability and willingness to comply with study procedures (e.g. stool collections) for the entire length of the study.
* Willing to provide consent/assent for the collection of stool samples.

Exclusion Criteria:

* Allergy to resistant starch or excipients.
* Co-existing diagnosis with diabetes mellitus.
* Treatment with another investigational drug or intervention throughout the study.
* Current drug or alcohol dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of an individual or legal guardian to give written informed consent.
* Requirement for antibiotic therapy as part of standard Crohn's Disease therapy (i.e. those patients with penetrating disease as manifested by intra-abdominal abscess or perianal abscess).
* Requirement of oral antibiotics for other conditions (e.g. acne).
* Participant's microbiota does not produce butyrate in response to any of the assembled panel of resistant starch as measured through the Rapid Assay of an Individual's Microbiome (RapidAIM) evaluation following enrollment.
* Requirement of therapy other than oral corticosteroid / aminosalicylates for induction therapy.
* Patients diagnosed with Inflammatory Bowel Disease-Unclassified.
* Refusal to undergo follow-up colonoscopy as part of current clinical practice guidelines for Crohn's Disease standard of care.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Increased potential for butyrate production and its level at the mucosal luminal interface following ingestion of an individualized resistant starch as assessed by meta-omics analysis. | 5 ± 1 months
Sustained increased potential of butyrate production 6 months following cessation of the use of individualized resistant starch as assessed by meta-omics analysis of stools. | 12 ± 2 months
The percentage of eligible inflammatory bowel disease (IBD) patients who will enter a resistant starch-based ingestion trial. | Enrollment
  Threshold of interest will be 50%.
Compliance of resistant starch intake by patient report. | 5 ± 1 months
Compliance of resistant starch intake by product reconciliation. | 5 ± 1 months

SECONDARY OUTCOMES:
Change in microbiome composition of cases towards the microbiome of controls as assessed by meta-omics analysis. | 5 ± 1 months and 12 ± 2 months
Changes in mitochondrial function due to ingestion of resistant starch as assessed by host proteomics of biopsy sampling. | Enrollment, and 5 ± 1 months
Change in clinical disease activity as measured by the wPCDAI for Crohn's Disease, the PUCAI and Partial Mayo Score for Ulcerative Colitis, and the PGA for both Crohn's Disease and Ulcerative Colitis. | Enrollment, 5 ± 1 months, and 12 ± 2 months
  Weighted Pediatric Crohn's Disease Activity Index (wPCDAI) ranges from 0 to 125 points (<12.5 = remission, 12.5 to 40.0 = mild, >40.0 = moderate, >57.5 = severe). The Pediatric Ulcerative Colitis Activity Index (PUCAI) ranges from 0 to 85 points (<10 = remission, 10 to 34 = mild, 35 to 64= moderate, >65 = severe). Partial Mayo Score ranges from 0 to 9 points (0 to 1 = remission, 2 to 4 = mild, 5 to 6 = moderate, 7 to 9 = severe). The Physician Global Assessment (PGA) ranges from 0 to 3 points (0 = normal, 1 = mild, 2 = moderate, 3 = severe).
Changes in patient reported disability outcomes as measured by the IBD Disability Index Questionnaire. | Enrollment, 5 ± 1 months, and 12 ± 2 months
  The IBD disability index consists of 28 questions and a higher overall score is indicative of greater disability.
Changes in patient, parent/caregiver reported quality of life outcomes as measured by the IMPACT III Questionnaires. | Enrollment, 5 ± 1 months, and 12 ± 2 months
  The IMPACT III questionnaire (a health related quality of life questionnaire) consists of 35 questions and ranges in score from 0 to 231. A higher score represents a higher quality of life. The IMPACT III-P Questionnaire is to be completed by the caregiver/guardian with a higher score also representing a higher quality of life.
Changes in intestinal mucosal inflammation by measuring fecal calprotectin through stool samples. | Enrollment, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 8 months, 10 months, and 12 months
Change in endoscopic disease activity measured during colonoscopies using the SES-CD for Crohn's Disease and the Mayo Endoscopic Sub Score and UCEIS for Ulcerative Colitis. | Enrollment, and 5 ± 1 months
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) measures disease inflammation (0 to 2= inactive, 3 to 6 = mild, 7 to 15 = moderate, >16 = severe). Mayo Endoscopic Sub Scores range from 0 to 3, with 0 representing a normal mucosa or inactive disease and 3 representing severe activity (spontaneous bleeding and large ulcerations). The Ulcerative Colitis Endoscopic Index of Severity (UCEIS) ranges from 0 to 8 (0 to 1 = remission, 2 to 4 = mild, 5 to 6 = moderate, and 7 to 8 = severe).
Change in histological scoring of acute and chronic inflammation collected through biopsies during colonoscopies and assessed using Naini and Cortina score for Crohn's disease and the Robarts Histopathological Index (RHI) for Ulcerative Colitis. | Enrollment, and 5 ± 1 months
  The Naini and Cortina score ranges from 0 to 10 for ileitis and 0 to 17 for colitis. For ileitis, the histopathological support for having IBD is either low (score < 2), moderate (score is 3 to 4), or high (score ≥ 5). For colitis, the likelihood of having IBD is either low (≤3), moderate (score is 4 to 8), or high (score ≥ 9). The Robarts Histopathological Index score ranges from 0 to 33 with a higher score representing more severe inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: David Mack, MD, FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario; Alain Stintzi, PhD, Principal Investigator — University of Ottawa
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No